CLINICAL TRIAL: NCT06024213
Title: French, Prospective, Post-marketing Study to Describe the Use, Detection Performance and Safety Profile of Infracyanine® (Indocyanine Green) for Breast Cancer Patients Undergoing a Sentinel Lymph Node (SLN) Biopsy.
Brief Title: A French Observational Study of Indocyanine Green for Patients With Breast Cancer Having a Sentinel Lymph Node Biopsy.
Acronym: OASIS
Status: Completed | Type: Observational
Sponsor: BTG International Inc. (Other)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: PR024-CLN-pro101
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
Keywords: sentinel lymph node biopsy; indocyanine green biopsy; fluorescence blue dye; technetium99
MeSH Terms: conditions — Breast Neoplasms | interventions — Indocyanine Green; Methylene Blue; Technetium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Sentinel lymph node identification — Intervention description: Intraoperative identification of sentinel lymph node
Drug: indocyanine green — Intervention description: indocyanine green (5 to 10 mg [ie, 2 to 4 mL of a 2.5 mg/mL solution]) administered by periareolar or peritumoural route
Drug: methylene blue — 1%), 2-5 mL administered by periareolar or peritumoural route
Drug: Technetium (99mTc) — (99mTc, 0.2 - 0.4 mCi in 0.4 mL administered by periareolar or peritumoural route

SUMMARY:
This prospective, observational study will evaluate the patient-based sentinel lymph node detection rate when using the Infracyanine® (indocyanine green) dye technique in patients undergoing surgery for breast cancer.

The study will describe the demographic, clinical, and tumour characteristics of patients with breast cancer undergoing surgery.

The study will describe the characteristics of how the indocyanine green dye technique is used including the dose and volume of dye used, the number and type of injection sites used to give the dye, the equipment used to detect the dye and locate the sentinel lymph node, and whether indocyanine green is used on its own or with other dyes (blue dye and/or 99mTechnetium dye).

The study will evaluate the characteristics of sentinel lymph node biopsy procedures performed using indocyanine green dye including the number of biopsies performed, the time taken to detect the sentinel lymph node and perform the biopsy, and how many sentinel lymph nodes are detected using indocyanine green dye, blue dye, and 99mTechnetium dye.

The study will also assess the safety of using indocyanine green dye for 6 weeks following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged ≥18 years
* Undergoing breast cancer surgery with an indication for sentinel lymph node biopsy
* Receiving Infracyanine® (indocyanine green; alone or in combination with blue dye or 99mTc) for intraoperative identification of sentinel lymph node according to the Summary of Product Characteristics

Exclusion Criteria:

* Male
* Pregnant or nursing female
* Previous allergy to indocyanine green or to any excipients
* Already included in a surgical trial
* Patient opposed to collection and processing of their data

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at French hospitals involved in the management of female patients with breast cancer where indocyanine green is used in routine practice. Patients will be enrolled from approximately 5 sites in metropolitan France.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Sentinel lymph node detection rate | Time of Surgery
  Rate of detection of at least one sentinel lymph node by indocyanine green

SECONDARY OUTCOMES:
Age | At visit 1 (pre-operative consultation)
  Patient age
Height | At visit 1 (pre-operative consultation)
  Patient height
Weight | At visit 1 (pre-operative consultation)
  Patient weight
BMI | At visit 1 (pre-operative consultation)
  Patient BMI
Comorbidities | At visit 1 (pre-operative consultation)
  Comorbidities of interest
Menopause status | At visit 1 (pre-operative consultation)
  Menopause status
Prior excisional surgery | At visit 1 (pre-operative consultation)
  Prior excisional surgery on the breast
Surgery type planned | At visit 1 (pre-operative consultation)
  Type of breast surgery planned
Tumour size | At visit 1 (pre-operative consultation)
  Tumour size
Tumour grade | At visit 1 (pre-operative consultation)
  Tumour grade
Tumour stage | At visit 1 (pre-operative consultation)
  Tumour stage
Histological type | At visit 1 (pre-operative consultation)
  Tumour histological type
Hormone receptor status | At visit 1 (pre-operative consultation)
  Tumour hormone receptor status (estrogen receptors, progesterone receptors, and HER2 status)
Tumour laterality | At visit 1 (pre-operative consultation)
  Tumour laterality
Tumour quadrant | At visit 1 (pre-operative consultation)
  Tumour quadrant
Detection method | Time of surgery
  Method used to detect sentinel lymph node (indocyanine green alone or in combination with blue dye or 99mTc)
Indocyanine green dose | Time of surgery
  Dose of indocyanine green
Indocyanine green volume | Time of surgery
  Volume of indocyanine green
Injection site | Time of surgery
  Description of injection site
Number of injection sites | Time of surgery
  Number of injection sites
Route of injection | Time of surgery
  Route of injection (periareolar or peritumoural)
Detection equipment | Time of surgery
  Equipment used for detection of sentinel lymph node
Number of sentinel lymph node biopsies performed | Time of surgery
  Number of sentinel lymph node biopsies performed
Time from injection to visualization | Time of surgery
  Time from injection to visualization of first sentinel lymph node
Time from injection to end of biopsy | Time of surgery
  Time from injection to end of biopsy procedure
Number of sentinel lymph nodes detected | Time of surgery
  Number of sentinel lymph nodes detected (by all detection methods) per patient
Number of sentinel lymph nodes detected - indocyanine green | Time of surgery
  Number of sentinel lymph nodes detected (by indocyanine green) per patient
Number of sentinel lymph nodes detected - blue dye | Time of surgery
  Number of sentinel lymph nodes detected (by blue dye) per patient
Number of sentinel lymph nodes detected - 99mTc | Time of surgery
  Number of sentinel lymph nodes detected (by 99mTc) per patient
Adverse events | From time of surgery up to 6 weeks post-surgery
  Number, frequency, grade, and outcomes of adverse events related to indocyanine green, using CTCAE v5 criteria/MedDRA
Serious adverse events | From time of surgery up to 6 weeks post-surgery
  Number frequency, and outcomes of serious adverse events related to indocyanine green, using CTCAE v5 criteria/MedDRA
Changes in vital signs | From time of surgery up to 6 weeks post-surgery
  Number of observed clinically significant changes in blood pressure, pulse rate, and respiratory rate

OTHER OUTCOMES:
Sentinel lymph node detection rate by obesity status | Time of surgery
  Rate of detection of at least one sentinel lymph node by indocyanine green in obese (BMI ≥30 kg/m2) vs non-obese (BMI ≤30 kg/m2) patients
Sentinel lymph node detection rate in early-stage breast cancer | Time of surgery
  Rate of detection of at least one sentinel lymph node by indocyanine green in patients with stage 1A, 1B, or 2A breast cancer
Sentinel lymph node detection rate by indocyanine green dose | Time of surgery
  Rate of detection of at least one sentinel lymph node by indocyanine green for patients receiving 5 mg dose vs 10 mg dose
Sentinel lymph node detection rate by injection route | Time of surgery
  Rate of detection of at least one sentinel lymph node by indocyanine green for patients injected via periareolar vs peritumoural vs subcutaneous route

CONTACTS AND LOCATIONS:
Overall Officials: Céline Chauleur, MD, Study Chair — CHU de Saint-Etienne
Locations (6):
- France (6):
  - CH Annecy-Genevois, Annecy, Epagny Metz-Tessy, Haute-Savoie
  - Institut Bergonié, Bordeaux, Gironde
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHU de Lille, Lille, Nord
  - CHU de Saint-Etienne, Saint-Étienne-de-Montluc, Pays de la Loire Region
  - Hôpital Européen Georges-Pompidou Paris, Paris, Île-de-France Region

REFERENCES:
- [Background] Vermersch C, Raia-Barjat T, Chapelle C, Lima S, Chauleur C. Randomized comparison between indocyanine green fluorescence plus 99mtechnetium and 99mtechnetium alone methods for sentinel lymph node biopsy in breast cancer. Sci Rep. 2019 May 6;9(1):6943. doi: 10.1038/s41598-019-43473-3. PMID 31061432
- [Background] Guo J, Yang H, Wang S, Cao Y, Liu M, Xie F, Liu P, Zhou B, Tong F, Cheng L, Liu H, Wang S. Comparison of sentinel lymph node biopsy guided by indocyanine green, blue dye, and their combination in breast cancer patients: a prospective cohort study. World J Surg Oncol. 2017 Nov 2;15(1):196. doi: 10.1186/s12957-017-1264-7. PMID 29096643
- [Background] Kitai T, Inomoto T, Miwa M, Shikayama T. Fluorescence navigation with indocyanine green for detecting sentinel lymph nodes in breast cancer. Breast Cancer. 2005;12(3):211-5. doi: 10.2325/jbcs.12.211. PMID 16110291
- [Background] Sugie T, Kinoshita T, Masuda N, Sawada T, Yamauchi A, Kuroi K, Taguchi T, Bando H, Yamashiro H, Lee T, Shinkura N, Kato H, Ikeda T, Yoshimura K, Ueyama H, Toi M. Evaluation of the Clinical Utility of the ICG Fluorescence Method Compared with the Radioisotope Method for Sentinel Lymph Node Biopsy in Breast Cancer. Ann Surg Oncol. 2016 Jan;23(1):44-50. doi: 10.1245/s10434-015-4809-4. Epub 2015 Aug 15. PMID 26275781